CLINICAL TRIAL: NCT01189877
Title: Characterization of Rectal Cancer Hypoxia Using pO2 Histography and Immunohistochemistry for Hypoxia-Related Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-121
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Rectal Cancer
Keywords: Direct pO2 Measurements; 10-121
MeSH Terms: conditions — Rectal Neoplasms

ARMS (1):
- pO2 measurements (Experimental): In patients meeting eligibility requirements outlined below, comparisons will be made between direct pO2 measurements using a tissue hypoximeter and IHC-assessed expression of hypoxia related proteins (HIF-1α, VEGF, CA IX and GLUT-1) in both normal and tumor tissue.
  Interventions: Procedure: Eppendorf hypoximeter

INTERVENTIONS:
Procedure: Eppendorf hypoximeter — Patients consented to the protocol will proceed to their surgery date without any change in the standard preoperative period. After arriving in the operating room, the patient will undergo intravenous general anesthesia (or spinal/epidural anesthesia) by the anesthesiologist and will receive 40% oxygen. At this time, the principal investigator (along with the assistance of the operating surgeon and a member of the Department of Medical Physics) will use the Eppendorf hypoximeter to gather pO2 measurements. We anticipate that this will add no more than fifteen minutes to the planned procedure. Once the measurements are collected, the anesthesia will be adjusted as appropriate for the surgery and the procedure will continue as usual.

SUMMARY:
The purpose of this study is to see if the cells in rectal cancer are oxygen-starved, or hypoxic. We know that as cancers grow bigger, parts of them are cut off from the oxygen supply and they become hypoxic, basically, lacking oxygen. Research has shown that cells that are oxygen-starved respond differently to treatment such as chemotherapy and radiation when compared to cells that are oxygen rich.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum. If a biopsy was taken at an outside hospital, the slides and diagnosis will be reviewed and confirmed by a pathologist at MSKCC.
* Mid to distal rectal tumors not requiring pre-op radiation or chemotherapy
* Age ≥ 18
* Age < 90
* Karnofsky performance status ≥ 60
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Current pregnancy
* Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Measure pO2 in rectal cancers | 2 years
  Measure pO2 in rectal cancers

SECONDARY OUTCOMES:
Correlate immunohistochemical analysis of endogenous markers of hypoxia | 2 years
  with direct tumor hypoximetry in tumor and normal tissue.

CONTACTS AND LOCATIONS:
Overall Officials: José Guillem, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm